CLINICAL TRIAL: NCT01301430
Title: Phase I/IIa Study of Intratumoral/Intracerebral or Intravenous/Intracerebral Administration of Parvovirus H-1 (ParvOryx) in Patients With Progressive Primary or Recurrent Glioblastoma Multiforme.
Brief Title: Parvovirus H-1 (ParvOryx) in Patients With Progressive Primary or Recurrent Glioblastoma Multiforme.
Acronym: ParvOryx01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oryx GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ParvOryx01
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2015-03

CONDITIONS: Glioblastoma Multiforme
Keywords: Progressive glioblastoma multiforme; Recurrent glioblastoma multiforme; Oncolytic virus
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- H-1 parvovirus (H-1PV) (Experimental)
  Interventions: Drug: H-1PV

INTERVENTIONS:
Drug: H-1PV — H-1PV administered at three increasing doses either intratumorally or intravenously and then 10 days after the first administration intracerebrally (into the walls of tumor resection cavity).
  Other Names: ParvOryx (brand name of H-1PV)

SUMMARY:
Investigation on safety, tolerability and efficacy of H-1 parvovirus (H-1PV) in subjects suffering from glioblastoma multiforme.

DETAILED DESCRIPTION:
Investigation on safety, tolerability and efficacy of H-1 parvovirus (H-1PV) in subjects suffering from glioblastoma multiforme.

H-1PV will primarily be administered either intratumoral or intravenously. Ten days thereafter a complete or a subtotal tumor resection with a subsequent administration of H-1PV into the walls of the resection cavity will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Age over or equal to 18 years old,
* Diagnosis of glioblastoma multiforme,
* Written informed consent,
* Recurrent or progressive disease despite previous radio- and/or chemotherapy,
* Indication for complete or subtotal tumor resection,
* Life expectancy of at least 3 months,
* Consent for sampling and investigation of biological specimens,
* Karnofsky Performance Score over or equal to 60,
* Adequate seizure control,
* Adequate bone marrow function: neutrophils > 1.5 x 10exp9/L, platelets > 100 x 10exp9/L, hemoglobin > 9.0 g/dL,
* Adequate liver function: Bilirubin < 2.0 g/dL, ASAT, ALAT, AP, GGT < 3 x ULN,
* Adequate renal function: Creatinine < 1.8 g/dL,
* Adequate blood clotting: aPTT < 35 sec, INR < 1.2,
* Negative serology for HIV, HBV and HCV,
* Negative Beta-HCG test in women of childbearing potential,
* Commitment to use adequate contraception (in both genders) for up to six months after study entry,
* Commitment to omit exposure to infants < 18 months of age or immunocompromised individuals for up to 28 day after first administration of IMP.

Exclusion Criteria:

* Multifocal disease,
* Evidence of distant tumor metastases,
* Contraindications for MRI,
* Active infection within 5 days prior to the study inclusion,
* Chemotherapy within 4 weeks prior to the study inclusion,
* Radiotherapy within 6 weeks prior to the study inclusion,
* Participation in another interventional trial within the last 30 days,
* Treatment with antiangiogenic substances within 21 days prior to therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 28 days after the first administration of the IMP
  Parameters for assessment of safety and tolerability:
  * physical/neurological examinations (pathological findings as quality and quantity)
  * adverse events (quality and quantity per dose level)
  * vital signs, ECG, laboratory parameters (pathological findings as quality and quantity, for laboratory parameters: descriptive statistics)
  * viral shedding and viral specific antibodies (quantity depicted over time)

SECONDARY OUTCOMES:
Efficacy (treatment response) | Up to 6 months after the first administration of the IMP
  Parameters for evaluation of efficacy:
  * Progression free survival (PFS) based on modified RECIST-criteria depicted as Kaplan-Meier curve
  * Overall survival (OS) depicted as Kaplan-Meier curve

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Unterberg, Prof. Dr., Principal Investigator — Department of Neurosurgery, University Hospital Heidelberg; Bernard Huber, Dr., Study Director — Oryx GmbH & Co. KG
Locations (1):
- Department of Neurosurgery, University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Geletneky K, Huesing J, Rommelaere J, Schlehofer JR, Leuchs B, Dahm M, Krebs O, von Knebel Doeberitz M, Huber B, Hajda J. Phase I/IIa study of intratumoral/intracerebral or intravenous/intracerebral administration of Parvovirus H-1 (ParvOryx) in patients with progressive primary or recurrent glioblastoma multiforme: ParvOryx01 protocol. BMC Cancer. 2012 Mar 21;12:99. doi: 10.1186/1471-2407-12-99. PMID 22436661
- [Background] Geletneky K, Leoni AL, Pohlmeyer-Esch G, Loebhard S, Baetz A, Leuchs B, Roscher M, Hoefer C, Jochims K, Dahm M, Huber B, Rommelaere J, Krebs O, Hajda J. Pathology, organ distribution, and immune response after single and repeated intravenous injection of rats with clinical-grade parvovirus H1. Comp Med. 2015 Feb;65(1):23-35. PMID 25730754
- [Background] Geletneky K, Leoni AL, Pohlmeyer-Esch G, Loebhard S, Leuchs B, Hoefer C, Jochims K, Dahm M, Huber B, Rommelaere J, Krebs O, Hajda J. Bioavailability, biodistribution, and CNS toxicity of clinical-grade parvovirus H1 after intravenous and intracerebral injection in rats. Comp Med. 2015 Feb;65(1):36-45. PMID 25730755
- [Background] Geletneky K, Hajda J, Angelova AL, Leuchs B, Capper D, Bartsch AJ, Neumann JO, Schoning T, Husing J, Beelte B, Kiprianova I, Roscher M, Bhat R, von Deimling A, Bruck W, Just A, Frehtman V, Lobhard S, Terletskaia-Ladwig E, Fry J, Jochims K, Daniel V, Krebs O, Dahm M, Huber B, Unterberg A, Rommelaere J. Oncolytic H-1 Parvovirus Shows Safety and Signs of Immunogenic Activity in a First Phase I/IIa Glioblastoma Trial. Mol Ther. 2017 Dec 6;25(12):2620-2634. doi: 10.1016/j.ymthe.2017.08.016. Epub 2017 Aug 24. PMID 28967558